CLINICAL TRIAL: NCT06153498
Title: A Randomized Study of the PK/PD Properties and Safety of Remazolam Besylate for Injection in ICU Patients With Impaired Renal Function
Brief Title: PK/PD Properties and Safety of Remazolam Besylate for Injection in ICU Patients With Impaired Renal Function
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Collaborators: Yichang Humanwell Pharmaceutical Co., Ltd., China (Industry)
Responsible Party: Principal Investigator, Xiaobo Yang, MD, MD, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: WHUICU202203
Record Dates: First submitted 2023-11-23; First posted 2023-12-01 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Mechanically Ventilated Patients

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normal renal function group (Experimental)
  Interventions: Drug: Remimazolam besylate
- Renal injury group (Experimental)
  Interventions: Drug: Remimazolam besylate

INTERVENTIONS:
Drug: Remimazolam besylate — After a loading dose of 0.05mg/kg, a maintaining dose of 0.2mg/kg/h is given; It is recommended to adjust the infusion rate of Remazolam besylate for injection at a amplitude of 0.05mg/kg/h, mainly based on the RASS score of the subjects (the adjustment range is 0-1.0 mg/kg/h, and the maximum infusion rate is not more than 1.0mg/kg/h) until the subjects reach the optimal sedation level (-3≤RASS≤0).

SUMMARY:
Pharmacokinetic/pharmacodynamic profiles of remazolam besylate were compared in patients with impaired and normal renal function in the ICU, and safety was assessed by recording hemodynamic parameters and adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) ≥18 and ≤ 30 kg/m2
* Being Intubated and mechanically ventilated ≤48 hours before enrollment and expected to be on a ventilator for at least 6 hours
* Requirement for light to moderate sedation (a Richmond agitation-sedation scale score of -2 to 1) Patients with impaired renal function were defined as having a glomerular filtration rate of 30 to 89 ml/min/1.73m2. Patients with normal renal function were defined as having a glomerular filtration rate of 90 to 120 ml/min/1.73m2

Exclusion Criteria:

* Refusal to be included
* Allergy or unsuitability to any composition of study drugs or remifentanil
* Living expectancy less than 48 hours
* Myasthenia gravis
* Status asthmaticus
* Abdominal compartment syndrome
* Serious hepatic dysfunction (CTP 10-15);
* Chronic kidney disease with glomerular filtration rate (GFR) < 29 ml/ min/1.73m2
* Mean blood pressure less than 65 mm Hg or the need for a continuous infusion of norepinephrine at ≥0.5 ug/kg/min to maintain Mean blood pressure ≥ 65 mm Hg
* Possible requirement for surgery or bedside tracheostomy in 24 hours
* Possible requirement for renal replacement therapy in 24 hours
* Acute severe neurological disorder and any other condition interfering with sedation assessment
* Abuse of controlled substances or alcohol
* Pregnancy or lactation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-11-04 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Cmax | Within 24 hours while receiving the study drug
  peak plasma concentration
The area under the plasma drug concentration-time curve | Within 24 hours while receiving the study drug
  The area under the plasma drug concentration-time curve (AUC)
t1/2 | Within 24 hours while receiving the study drug
  half-life

SECONDARY OUTCOMES:
The percentage of time in the target sedation range without rescue sedation | Within 24 hours while receiving the study drug
  The percentage of time in the target sedation range without rescue sedation
The number and severity of treatment emergent adverse events (TEAEs) | Within 24 hours while receiving the study drug
  The number and severity of treatment emergent adverse events (TEAEs)

CONTACTS AND LOCATIONS:
Locations (1):
- Wuhan Union Hospital, Wuhan, Hubei, China